CLINICAL TRIAL: NCT02088398
Title: Open-Label, Randomized, Single Dose, 3-Period Crossover to Evaluate the Relative Bioavailability and Food-Effect on Pharmacokinetics of Alternative 10 mg/mL Liquid Formulation ACY-1215 (Ricolinostat) in Healthy Subjects
Brief Title: Alternative 10 mg/mL Liquid Formulation of ACY 1215 (Ricolinostat) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acetylon Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ACE-HV-100
Record Dates: First submitted 2014-03-05; First posted 2014-03-17 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: relative bioavailability; food-effect
MeSH Terms: interventions — ricolinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 160 mg ACY-1215 CLF (20 mg/mL) fed (Experimental): • Treatment A: a single dose of 160 mg ACY-1215 CLF (20 mg/mL) in the fed state
  Interventions: Drug: ACY-1215
- 120 mg ACY-1215 ALF (10 mg/mL) fed (Experimental): • Treatment B: a single dose of 120 mg ACY-1215 ALF (10 mg/mL) in the fed state
  Interventions: Drug: ACY-1215
- 120 mg ACY-1215 ALF (10 mg/mL) fasted (Experimental): • Treatment C: a single dose of 120 mg ACY-1215 ALF (10 mg/mL)
  Interventions: Drug: ACY-1215

INTERVENTIONS:
Drug: ACY-1215

SUMMARY:
This study will be an open-label, randomized, single dose, 3-period crossover PK study. This study will comprise 3 treatment periods with a 4-day washout between periods. On Day -1, subjects will be randomized to 1 of 6 treatment sequences. On Days 1, 5, and 9, subjects will be administered Treatment A, B, or C according to the randomization schedule.

* Treatment A: a single dose of 160 mg ACY-1215 CLF (20 mg/mL) in the fed state
* Treatment B: a single dose of 120 mg ACY-1215 ALF (10 mg/mL) in the fed state
* Treatment C: a single dose of 120 mg ACY-1215 ALF (10 mg/mL) in the fasted state

DETAILED DESCRIPTION:
Subjects will be confined to the Clinical Research Unit (CRU) from the time of Check-in (Day -1) to Day 10. Predose blood and urine samples will be obtained prior to each ACY-1215 administration. Following administration of ACY-1215 in each period, blood and urine samples will be collected at specified timepoints or intervals through 24 hours postdose for the determination of the PK of a single oral dose of ACY-1215. Subjects will be discharged from the CRU on Day 10, following the completion of the last PK collection and successful completion and evaluation of discharge safety tests. Subjects will return to the clinic for a Follow-up visit 5 to 7 days after the last dose of ACY-1215 (Days 14 to 16) for additional safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age, inclusive
* BMI range 18.5 to 32.0 kg/m2
* in good health, as determined by no clinically significant findings from medical history, 12-lead ECG, vital signs
* clinical laboratory evaluations, CBC, coagulation, and UA
* negative test for selected drugs of abuse
* negative hepatitis panel and negative HIV antibody
* females of non-childbearing potential as outlined in protocol
* males either be sterile or agree to use contraception as outlined in protocol

Exclusion Criteria:

* significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* history of Gilbert's Syndrome or suspicion of Gilbert's Syndrome
* abnormality in the 12-lead ECG (e.g. QTcF of >450 msec, a history of a prolonged QTc-interval or Brugada syndrome)
* history of alcoholism or drug addiction within 1 year prior
* participation in any other investigational study drug trial in which receipt of an investigational study drug as outlined in protocol
* use of any prescription medications/products within 14 days (30 days for cytochrome P450 [CYP]-inducing or inhibiting products as outlined in protocol)
* use of any over-the-counter, nonprescription preparations within 14 days
* use of any tobacco or nicotine-containing products within 6 months and during study;
* poor peripheral venous access
* donation of blood from 30 days prior to Screening through the Follow-up visit
* any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Zero to Last Time - AUC0-last | 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hr post first dose

SECONDARY OUTCOMES:
Safety and tolerability parameters | Day 1 (first dose of ACY-1215) to Day 16
  Changes from baseline in clinical laboratory assessments, vital signs, electrocardiogram values, and physical exam. This includes collection of adverse events and the collection of concomitant medications.
Area Under the Curve From Time Zero to Extrapolated Infinite Time | 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hr post first dose
Maximum Observed Plasma Concentration (Cmax) | 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hr post first dose
Plasma Decay Half-Life | 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hr post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, M.D., Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Incorporated, Madison, Wisconsin, United States